CLINICAL TRIAL: NCT04455646
Title: Combining H1-Coil Deep Transcranial Magnetic Stimulation (dTMS) and App-guided CBT in Subjects With Major Depression Disorder (MDD)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Brainsway (Industry)
Responsible Party: Sponsor
Other Study IDs: 101
Record Dates: First submitted 2020-06-29; First posted 2020-07-02 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-06

CONDITIONS: Data Collection for Facilitation of Machine Learning Algorithm for Personalized Treatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Behavioral: CBT-based, mobile-delivered, intervention platform — App of this platform have been shown to be associated with reduced psychopathology symptoms,including depressive symptoms, following treatment (i.e., relapse prevention). GGDE, which was specifically designed to address MDD related maladaptive beliefs and symptoms,includes different CBT-based intervention modules (nine active and one sham), as well as means for data collection and response monitoring. The active treatment modules will differ in the proportion of adaptive vs. maladaptive statements and the emphasis on particular content (e.g loneliness vs. hopelessness).

SUMMARY:
A naturalistic study design, in which dTMS patients will be randomized to get a free add-on CBT treatment. The dTMS procedure will include treatment as usual, and participants will use the app from post randomization (Pre-treatment is defined as measures from the first three days of treatment) to the end of dTMS treatment (Post-treatment which is defined as measures from after twenty TMS sessions over a minimum of four weeks), and for an additional three months of FU (FU).

DETAILED DESCRIPTION:
Participants will be recruited from those attending dTMS clinics around the world (i.e.,naturalistic study design), and consenting individuals (in person consent done in the clinic on paper) will be given a random user code. This code will be specific for their version of the app, and the only link between their signature and the code will remain at the site for auditing purposes. Participants will undergo treatment as usual of dTMS and will use GGDE twice a day. Participants will be asked to complete demographic and clinical questionnaires via the GGDE app, and relevant clinical questionnaires will be re-administered following treatment and during FU. The initial and all following dTMS sessions will involve patients going through the stimulation procedure (The operator will record stimulation variables such as individual patient's intensity of stimulation and coil location into GGDE) followed by 5 min of GGDE use. The patient will indicate which statements (in that session) were most relevant and challenging to them, which will be followed by a pre-prepared psycho-education paragraph about the specific maladaptive belief addressed by the app that day. The patient will then be prompted to use the app one more time at home during the same day. Patient will continue similar use during FU, with two GGDE usage each day. The naturalistic design will allow the accumulation of large quantities of data in a short period of time, aiming to optimize GGDE using machine learning. Importantly, GGDE will allow the random allocation of users to different GGDE modules of the app (i.e., similar app versions with changes in specific parameters related to different depressive traits). One out of the ten modules used in this trial will include neutral (placebo) stimuli requiring the user to respond to plus/minus signs rather than MDD relevant statements.

ELIGIBILITY:
Inclusion Criteria:

* Adult outpatients accepted to treatment as usual dTMS with a Primary DSM-V diagnosis of Major Depression, single or recurrent episode
* Capable and willing to provide informed consent
* In a possession of a Smartphone capable of running the GGDE app.
* Able to adhere to the treatment schedule.

Exclusion Criteria:

Investigators, site personnel directly affiliated with this study, and their immediate families (immediate family is defined as a spouse, parent, child or sibling, whether by birth or legal adoption).

-

Ages: 22 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The intention is to enroll at least 540 patients diagnosed with MDD who were accepted into dTMS treatment for depression. The patients will be of all racial, ethnic and gender categories. The course of illness histories will be based upon patient reporting through the GGDE app. Patients who are unlikely to show response based on the literature to date (presence of psychosis, co-morbid and prominent anxiety disorder or substance abuse, personality disorder or dysthymia) will not be asked to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 540 (Estimated)
Dates: Start 2019-08-26 (Actual); Primary Completion 2021-08-26 (Estimated); Study Completion 2021-08-26 (Estimated)

PRIMARY OUTCOMES:
Patient Patient Health Questionnaire (PHQ) Patient Health Questionnaire (PHQ) Patient Health Questionnaire (PHQ) Health Questionnaire (PHQ) | 1 year
  The change from Pre- to Post-treatment in the Patient Health Questionnaire (PHQ) scores from baseline to endpoint.

SECONDARY OUTCOMES:
Patient Patient Health Questionnaire (PHQ) | 1 year
  Response rate (50% reduction from Pre-treatment of the PHQ score), where the rate refers to the percentage of patients in response at Post-treatment.
  * Remission rate (PHQ<5; [1]), where the rate refers to the percentage of patients in remission at Post-treatment,
  * Response rate, Remission rate, and the change from Pre-treatment to FU in the PHQ score.

CONTACTS AND LOCATIONS:
Locations (22):
- United States (22):
  - Kadima Neuropsychiatry, San Diego, California
  - Advanced Mental Health Care Inc. - Juno Beach, Juno Beach, Florida
  - Advanced Mental Health Care Inc. - Palm Beach, Palm Beach, Florida
  - Advanced Mental Health Care Inc. - Royal Palm Beach, Royal Palm Beach, Florida
  - Greenbrook - Annapolis, Annapolis, Maryland
  - Greenbrook - Columbia, Columbia, Maryland
  - Greenbrook - Frederick, Frederick, Maryland
  - Greenbrook - Glen Burnie, Glen Burnie, Maryland
  - Greenbrook - Greenbelt, Greenbelt, Maryland
  - Greenbrook - Kensington, Kensington, Maryland
  - Greenbrook - Olney, Olney, Maryland
  - Greenbrook - Rockville, Rockville, Maryland
  - Greenbrook - O'Fallon, O'Fallon, Missouri
  - Greenbrook - Tesson Ferry, St Louis, Missouri
  - Greenbrook - Creve Coeur, St Louis, Missouri
  - Greenbrook - Chapel Hill, Chapel Hill, North Carolina
  - Greenbrook - Greensboro, Greensboro, North Carolina
  - Greenbrook - Matthews, Matthews, North Carolina
  - Greenbrook - Raleigh, Raleigh, North Carolina
  - Greenbrook - Glen Allen, Glen Allen, Virginia
  - Greenbrook TMS NeuroHealth Centers, McLean, Virginia
  - Greenbook - Newport News, Newport News, Virginia

IPD SHARING:
Plan to Share IPD: No